CLINICAL TRIAL: NCT06192576
Title: A Prospective Observational Study to Assess the Long-term Safety and Immunogenicity of Olipudase Alfa Therapy During Routine Clinical Care in Pediatric Patients Less Than 2 Years of Age With Acid Sphingomyelinase Deficiency
Brief Title: A Real-world Long-term Safety and Immunogenicity Study of Olipudase Alfa Therapy in Pediatric Patients Less Than 2 Years of Age With Acid Sphingomyelinase Deficiency (ASMD)
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Pulse Infoframe Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18020; U1111-1294-8169 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Niemann-Pick Diseases; Acid Sphingomyelinase Deficiency
MeSH Terms: conditions — Niemann-Pick Diseases | interventions — olipudase alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Olipudase alfa arm
  Interventions: Drug: Olipudase alfa

INTERVENTIONS:
Drug: Olipudase alfa — This study will not administer any treatment, only observe the treatment as prescribed in real-world clinical practice.
  Other Names: Xenpozyme®

SUMMARY:
US, multicenter, cohort, open label observational study with primary data collection. Ancillary protocol-specified procedures to address the study objectives (eg, assessment of ADA) may be considered outside the standard of care for acid sphingomyelinase deficiency (ASMD), but the study methodology remains non-interventional, as the additional collection of data from participants will not dictate treatment. The total overall study duration will be 5 years. The follow-up period will be a minimum of 1 year to a maximum of 3 years. The enrollment period will be up to 4 years, to allow a minimum of 1 year of follow-up for the last participant enrolled.

DETAILED DESCRIPTION:
This is a hybrid study design. Patients need not travel to existing study sites in order to enroll.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have ASMD type A/B or B and must be <2 years of age at the time of treatment initiation, OR ASMD type A (without age restriction).
* The participant must weigh ≥ 2 kg [The United States Prescribing Information (USPI)] for olipudase alfa specifies this minimum weight for infants receiving olipudase alfa).
* The participant must have documented ASMD, as determined in peripheral leukocytes, cultured fibroblasts, or lymphocytes and/or by genotype determination.
* Signed informed consent must be provided by the participant's parent(s)/legal guardian(s), including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. The signed ICF must be provided before any protocol-related procedures are performed.
* The participant is eligible to start olipudase alfa enzyme replacement therapy or has received the first dose (and no more) of olipudase alfa, and has retrievable clinical, laboratory, and ADA data.

Exclusion Criteria:

* The participant has received an investigational drug within 30 days or 5 drug half-lives before signature of the ICF and study enrollment.
* The participant is not suitable for participation for reasons determined by the Investigator, including medical or clinical conditions, or potential risk of noncompliance with study procedures.
* The participant is an immediate family member of employees of the study site or other individuals directly involved in study conduct, in conjunction with Section 1.61 of ICH-GCP Ordinance E6.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children under the age of 2 years with a documented ASMD diagnosis as shown by ASM deficiency in a cell-based assay (peripheral leukocytes, cultured fibroblasts, or lymphocytes) and/or by genotype determination will be considered for enrollment into this ASMD study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2029-01-02 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of cases in the exposed population with AEs, SAEs, and AESIs (including moderate/severe or recurrent hypersensitivity reactions and infusion-associated reactions) | Baseline to 3 years
Presence and titers of serum anti-olipudase alfa IgG anti-drug antibodies (ADA) (and IgE ADA in cases of moderate/severe or recurrent reactions) | Baseline to 3 years
Number of cases in the exposed population with abnormal laboratory test results and vital signs | Baseline to 3 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Ann and Robert H Lurie Children's Hospital of Chicago- Site Number: 001002, Chicago, Illinois
  - Children's Hospital Medical Center- Site Number: 001003, Cincinnati, Ohio
  - Nationwide Children's Hospital - PIN- Site Number : 1001-1, Columbus, Ohio
  - Pulse InfoFrame US Inc.- Site Number: 001001, Philadelphia, Pennsylvania
  - Dell Children's Medical Center- Site Number : 1001-2, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Register (healthie.net) — https://asmd.healthie.net/register